CLINICAL TRIAL: NCT01259011
Title: A Randomized Controlled Trial of SPIRIT: A Representational Intervention to Promote Preparation for End-of-Life Decision Making
Brief Title: A Representational Intervention to Promote Preparation for End-of-life Decision Making
Acronym: SPIRIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Mi-Kyung Song, PhD, RN, FAAN, Associate Professor, University of North Carolina, Chapel Hill
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 09-1190; R01NR011464 (NIH)
Record Dates: First submitted 2010-12-06; First posted 2010-12-13 (Estimated); Results first posted 2017-09-25 (Actual); Last update posted 2017-09-25 (Actual); Status verified 2017-07

CONDITIONS: End Stage Renal Disease
Keywords: end stage renal disease; dialysis; end of life decision making; surrogate psychological morbidities
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- control (No Intervention): Written information on advance directives and the patient's right to have an advance directive is provided to every patient on the first day of dialysis treatment by a social worker at the clinic. A social worker documents whether the patient has an advance directive, a surrogate decision maker, and/or a Do-Not-Resuscitate (DNR) Order on a Comprehensive Interdisciplinary Assessment form. The social worker encourages patients to complete an advance directive and addresses their questions about life-sustaining treatment options. If completed, the advance directive is placed in the medical record.
- SPIRIT intervention (Experimental): The SPIRIT intervention is a two-session, 1½ hour-long, structured intervention that is composed of six steps (assessing representations, identifying and exploring gaps and concerns, creating conditions for conceptual change, introducing replacement information, summarizing, and setting goals and planning), presented to both patient and surrogate by a trained nurse interventionist in a face-to-face interview format based on the representational approach.
  Interventions: Behavioral: the SPIRIT intervention

INTERVENTIONS:
Behavioral: the SPIRIT intervention — the SPIRIT intervention (Sharing the Patient's Illness Representation to Increase Trust) to improve discussions about end-of-life care between patients and their surrogate decision makers
  Arms: SPIRIT intervention

SUMMARY:
The proposed randomized controlled trial will test the SPIRIT (Sharing the Patient's Illness Representations to Increase Trust) intervention designed to improve discussions about end-of-life care between patients and their surrogate decision makers. Subjects will be 200 Caucasian and African-American patients with ESRD (end-stage renal disease) recruited from outpatient dialysis clinics and their chosen surrogate decision makers. We hypothesize that (1) SPIRIT will lead to significantly less patient decisional conflict and significantly greater dyad congruence and surrogate decision making confidence than the standard care control at 2, 6, and 12 months post-intervention and (2) SPIRIT will reduce surrogate decisional conflict and psychosocial morbidities at 2 weeks after the patient's hospitalization requiring surrogate decision making significantly more than the standard care control.

DETAILED DESCRIPTION:
Dialysis is central to survival for 450,000 Americans with end-stage renal disease (ESRD). Yet patients on dialysis have significant comorbidities and high mortality rates (24% annually). One out of four ESRD patient deaths occurs after a decision to stop dialysis. However, when persons have lost their decision capacity if there has been no prior discussion between the patient and surrogate regarding goals of care, the issue of whether to continue dialysis can pose an ethical impasse and cause profound psychological distress for surrogate decision makers. Using the representational approach to patient education, we developed and pilot tested the SPIRIT intervention (Sharing the Patient's Illness Representation to Increase Trust) to improve discussions about end-of-life care between patients and their surrogate decision makers. SPIRIT is a 6-step, 2-session, face-to-face intervention presented to both patient and surrogate by a trained interventionist in an interview format.

The proposed randomized controlled trial will test the effects of the SPIRIT intervention in improving preparedness for end-of-life decision making among ESRD patients and their surrogates and reducing surrogates' conflict during decision making and psychosocial morbidities. Subjects will be 200 Caucasian and African-American patients with ESRD recruited from outpatient dialysis clinics and their chosen surrogate decision makers. Preparedness outcomes (dyad congruence, patient decisional conflict, and surrogate decision making confidence) will be measured at 2, 6, and 12 months post-intervention. Surrogate decisional conflict and psychosocial morbidities (anxiety, depression, and post-traumatic distress symptoms) will be measured 2 weeks after the patient's hospitalization that required surrogate decision making. To compare the effects of SPIRIT to those of standard care on surrogates after the patient's death, psychosocial morbidities will be measured at 3 and 6 months after the patient's death. We will also explore the potential impact of race on intervention effects and examine mediators and moderators of the intervention effects.

ELIGIBILITY:
Inclusion Criteria:

for patients,

* self-identified Caucasian or African American;
* receiving either center-hemodialysis or home-peritoneal dialysis for at least 6 months prior to enrollment;
* availability of an individual chosen by the patient who can be present during the intervention as a surrogate decision maker;
* age 18 years or older;
* ability to participate in health care decisions as evidenced by less than 3 errors on the Short Portable Mental Status Questionnaire (SPMSQ), suggesting normal mental functioning;
* ability to read, write, and speak English.
* a CCI score of ≥6;
* hospitalization in the last 6 months, a CCI score of 5, including congestive heart failure (CHF).

for surrogates,

* age 18 years or older (to serve as a surrogate decision maker, the individual must be an adult);
* willingness to serve as the surrogate decision maker and participate in the intervention with the patient;
* ability to read, write, and speak English.

Exclusion Criteria:

-Patients who are too sick to participate in an hour-long interview, who require special care and assistance, who would not be able to care for their needs will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2010-03; Primary Completion 2014-02 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mi-Kyung Song, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina, Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Song MK, Ward SE, Fine JP, Hanson LC, Lin FC, Hladik GA, Hamilton JB, Bridgman JC. Advance care planning and end-of-life decision making in dialysis: a randomized controlled trial targeting patients and their surrogates. Am J Kidney Dis. 2015 Nov;66(5):813-22. doi: 10.1053/j.ajkd.2015.05.018. Epub 2015 Jun 30. PMID 26141307
- [Result] Song MK, Ward SE, Lin FC, Hamilton JB, Hanson LC, Hladik GA, Fine JP. Racial Differences in Outcomes of an Advance Care Planning Intervention for Dialysis Patients and Their Surrogates. J Palliat Med. 2016 Feb;19(2):134-42. doi: 10.1089/jpm.2015.0232. PMID 26840848
- [Result] Song MK, Ward SE, Hanson LC, Metzger M, Kim S. Determining Consistency of Surrogate Decisions and End-of-Life Care Received with Patient Goals-of-Care Preferences. J Palliat Med. 2016 Jun;19(6):610-6. doi: 10.1089/jpm.2015.0349. Epub 2016 Mar 16. PMID 26982909
- [Result] Song MK, Metzger M, Ward SE. Process and impact of an advance care planning intervention evaluated by bereaved surrogate decision-makers of dialysis patients. Palliat Med. 2017 Mar;31(3):267-274. doi: 10.1177/0269216316652012. Epub 2016 Jul 10. PMID 27272317
- [Derived] Song MK, Ward SE. The extent of informed decision-making about starting dialysis: does patients' age matter? J Nephrol. 2014 Oct;27(5):571-6. doi: 10.1007/s40620-014-0061-4. Epub 2014 Feb 12. PMID 24519843

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited between March 2010 and December 2012 from 20 outpatient dialysis centers in eight counties in North Carolina.
  A short battery of questions was used to help patients identify or confirm a previously designated surrogate. Patients and surrogates provided written consent.
Groups:
- Control: As required by Medicare and Medicaid programs (conditions for coverage for ESRD facilities), written information on advance directives and the patient's right to have an advance directive is provided to every patient on the first day of dialysis treatment by a social worker at the clinic. Also, the social worker documents whether the patient has an advance directive, a surrogate decision maker, and/or a Do-Not-Resuscitate (DNR) Order on a Comprehensive Interdisciplinary Assessment form. The social worker encourages patients to complete an advance directive and addresses their questions about life-sustaining treatment options. If completed, the advance directive is placed in the medical record.
Period: Main Study Period
Arm/Group | Control | SPIRIT Intervention
Started | 101 (101 dyads (=202 individuals)) | 109 (109 dyads (=218 individuals))
Completed | 101 | 109
Not Completed | 0 | 0
Period: After Patient Death
Arm/Group | Control | SPIRIT Intervention
Started | 17 (of 101 patient-surrogate dyads/pairs randomized, 17 surrogates of patients who died) | 28 (of 109 patient-surrogate dyads/pairs randomized, 28 surrogates of patients who died)
Completed | 17 | 28
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | SPIRIT Intervention | Total
Number analyzed (Participants) | 101 | 109 | 210
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.2 (11.1) | 61.1 (11.4) | 62.1 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 65 | 120
  Male | 46 | 44 | 90
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 69 | 72 | 141
  White | 32 | 37 | 69
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: patients]
  United States | 101 | 109 | 210

OUTCOME MEASURES:

1. Primary Outcome: Dyad Congruence
Description: patient and surrogate congruence on the goals of care
Time Frame: 2, 6, 12 months
Population: patients on dialysis and their surrogates
Measure: Number; unit: percentage of congruent dyads
Arm/Group | Control | SPIRIT Intervention
Number analyzed (Participants) | 101 | 109
percentage of congruent dyads | 48 | 64
Statistical Analysis 1: Comparison: Control vs SPIRIT Intervention; Test type: Superiority or Other; p < .05, Mixed Models Analysis; Odds Ratio (OR) = 1.9, 95% CI 2-sided [1.1 to 3.3]

2. Secondary Outcome: Change Over Time: Hospital Anxiety and Depression Scale Scores
Description: Hospital anxiety and depression (HADS) scores range from 0 to 21 with higher scores indicating greater symptom severity.
Time Frame: 2 Weeks, and at 3 and 6 months post death
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control | SPIRIT Intervention
Number analyzed (Participants) | 17 | 28
units on a scale
  Baseline HADS (Anxiety) | 6.1 (4.0) | 6.1 (4.2)
  2-Week F-Up HADS (Anxiety) | 6.6 (4.0) | 6.3 (2.6)
  3-Month F-Up HADS (Anxiety) | 6.4 (2.7) | 5.1 (2.6)
  6-Month F-Up HADS (Anxiety) | 6.6 (2.7) | 4.7 (3.4)
  Baseline HADS (Depression) | 3.1 (3.2) | 4.1 (3.1)
  2-Week F-Up HADS (Depression) | 6.4 (4.4) | 4.8 (3.2)
  3-Month F-Up HADS (Depression) | 5.9 (3.2) | 3.3 (3.1)
  6-Month F-Up HADS (Depression) | 5.9 (3.2) | 3.4 (2.8)
Statistical Analysis 1: Comparison: Control vs SPIRIT Intervention; Test type: Superiority; p = 0.12, Regression, Linear — HADS-anxiety; Slope = -1.2, 95% CI 2-sided [-2.8 to 0.3]
Statistical Analysis 2: Comparison: Control vs SPIRIT Intervention; Test type: Superiority; p < 0.05, Regression, Linear — HADS-depression; Slope = -2.2, 95% CI 2-sided [-4.2 to -0.3]

3. Secondary Outcome: Change Over Time: Post-traumatic Distress Symptom Score
Description: The Post-Traumatic Symptoms Scale-10 (PTSS-10) was used to assess the presence and intensity of PTSD symptoms during the preceding 7 days. This self-report scale consists of 10 statements that specifically mention symptoms related to PTSD criteria (e.g., sleep problems, nightmares, tension in the body, irritation, startle, etc.) rated on a 7-point Likert scale from 1 (Never/Rare) to 7 (Very often/Always). A total score (range 10 - 70) of > 35 is associated with a high probability that the person meets the diagnostic criteria for PTSD.
Time Frame: 2 weeks and 3 and 6 months after patient death
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control | SPIRIT Intervention
Number analyzed (Participants) | 17 | 28
units on a scale
  Baseline | 17.3 (8.1) | 20.2 (8.7)
  2-Week F-Up | 27.0 (14.0) | 23.6 (11.8)
  3-Month F-Up | 22.5 (8.3) | 19.3 (9.9)
  6-Month F-Up | 25.5 (12.4) | 20.3 (11.1)
Statistical Analysis 1: Comparison: Control vs SPIRIT Intervention; Test type: Superiority; p = 0.21, Regression, Linear; Slope = -4.0, 95% CI 2-sided [-10.2 to 2.2]

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 1 year
Arm/Group | Control | SPIRIT Intervention
All-Cause Mortality (participants affected / at risk) | 17/101 | 28/109
Serious Adverse Events (participants affected / at risk) | 0/101 | 0/109
Other Adverse Events (participants affected / at risk) | 0/101 | 0/109

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No